CLINICAL TRIAL: NCT00640978
Title: Phase II Study of Erlotinib and RAD001 (Everolimus) in Patients With Previously Treated Advanced Pancreatic Cancer
Brief Title: Erlotinib and RAD001 (Everolimus) in Patients With Previously Treated Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Significant Adverse Effects - Futility
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0666
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Advanced Pancreatic Cancer; Unresectable; Metastatic; RAD001; Everolimus; Erlotinib; OSI-774; Erlotinib Hydrochloride; Tarceva
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Everolimus; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib + RAD001 (Experimental): Erlotinib 150 mg orally daily for 28 Days + RAD001 (Everolimus) 30 mg orally weekly for 4 Weeks
  Interventions: Drug: RAD001; Drug: Erlotinib

INTERVENTIONS:
Drug: RAD001 — 30 mg orally weekly for 4 weeks
  Other Names: Everolimus
Drug: Erlotinib — 150 mg by mouth daily for 28 Days
  Other Names: Erlotinib Hydrochloride; OSI-774; Tarceva

SUMMARY:
The goal of this clinical research study is to learn if the combination of RAD001 and erlotinib hydrochloride can slow the growth of advanced pancreatic cancer. The safety of this drug combination will also be studied.

Primary Objectives:

-Determine the overall survival (OS) at 6 months of the combination of erlotinib and RAD001 in patients who have received previous treatment for advanced pancreatic cancer.

Secondary Objectives:

* Determine the progression-free survival (PFS).
* Determine the response rate (RR).

DETAILED DESCRIPTION:
The Study Drugs:

RAD001 is designed to stop cancer cells from multiplying. It may also stop the growth of new blood vessels that help tumor growth, which may cause the tumor cells to die.

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take erlotinib hydrochloride by mouth every day of each 28-day study "cycle". You should take erlotinib hydrochloride once a day in the morning with 1 cup (about 8 oz.) of water. Erlotinib hydrochloride should be taken at least 1 hour before or 2 hours after you have any food, vitamins, iron supplements, or other non-prescription drugs.

On Days 1, 8, 15, and 22 of each cycle, you will take RAD001 by mouth in the morning. You should either take the study drug on an empty stomach with 2 cups (about 16 oz.) of water or after a low-fat meal. You should not take the study drug after large fatty meals because fatty meals lower the amount of the study drug in your body. Some examples of a low-fat meal include cereal with fat-free milk, a low-fat muffin, toast, or a bagel with fat-free spread, or fruit salad.

On days when you take both RAD001 and erlotinib hydrochloride, RAD001 should be taken right before erlotinib hydrochloride.

If you experience intolerable side effects, you must call your doctor right away. The doctor may tell you to stop taking the study drugs or to take fewer pills. The study drugs may also be stopped completely, if your doctor thinks it is necessary.

Study Visits:

On Day 1 of every cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a performance status evaluation.
* Blood (about 2 tablespoons) and urine will for collected for routine tests. You should be fasting at the time of the blood draw. You should not eat or drink anything except water after midnight the night before.
* You will be asked about any drugs you may be taking or have taken since your last visit.

On Day 8 of Cycle 1, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 2 tablespoons) and urine will be collected for routine tests. You should be fasting at the time of the blood draw. You should not eat or drink anything except water after midnight the night before.
* You will be asked about any drugs you may be taking or have taken since your last visit.

At the end of every even cycle (Cycles 2, 4, 6, and so on), you will have a CT or MRI scan to check the status of the disease. The scans will be the same type that you had during screening.

Length of Study:

You may remain on study as long as you are benefitting. You will be taken off study early if the disease gets worse, you have intolerable side effects, or if your doctor decides that it is in your best interest to stop treatment.

End-of-Study Visit:

About 14 days after the last dose of study drug, you will have an end-of-study visit. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a performance status evaluation.
* Blood (about 2-3 tablespoons) and urine will be collected for routine tests. You should be fasting at the time of the blood draw. You should not eat or drink anything except water after midnight the night before.
* If you have not had them within the last 4 weeks, you will have a CT or MRI scan to check the status of the disease. The scans will be the same type that you had during screening.

Long-Term Follow-Up:

After you go off study, you will be asked how you are doing once a month for the first 6 months from the beginning of the study treatment. Then you will be asked how you are doing every 3 months from then on. This may be done either by phone contact or a clinic visit and will take about 15-30 minutes.

This is an investigational study. Erlotinib hydrochloride in combination with gemcitabine is commercially available and FDA approved for the treatment of pancreatic cancer. RAD001 is not FDA approved or commercially available. At this time, the combination of these drugs is only being used in research.

Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced pancreatic adenocarcinoma that is unresectable or metastatic.
* Patients must have received at least one prior chemotherapy regimen for unresectable/ metastatic disease. There is no limit to number of prior regimens. Prior erlotinib therapy is allowed.
* Minimum of two weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy. Patients must have recovered from the acute toxicities of any prior therapy to NIH-NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 </= Grade 1.
* Age >/= 18 years. Because no dosing or adverse event data are currently available on the use of erlotinib administered in combination with RAD001 in patients < 18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patients must have at least one measurable site of disease according to Response Evaluation Criteria In Solid Tumors (RECIST). This site must be outside a radiation field.
* Adequate hematologic, hepatic and renal parameters: leukocytes =/>3,000/ul, absolute neutrophil count =/>1,500/ul, platelets =/>100,000/ul, hemoglobin =/>9g/dL, total bilirubin </= 1.5 mg/dl, aspartate aminotransferase (AST) </=230 and alanine aminotransferase (ALT) </=280 IU/L for subjects with documented liver metastases; AST </=115 and ALT </=140 IU/L for subjects without evidence of liver metastases, creatinine </=1.5 mg/dl in males, </= 1.2 mg/dl in females.
* Women of childbearing potential (WOCBP) and men must agree to use adequate contraception prior to study entry for the duration of study treatment and 30 days after the end of treatment. WOCBP is defined as a woman who has not been naturally postmenopausal for at least 12 consecutive months or no previous surgical sterilization. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions and are therefore not considered effective for this study. WOCBP must provide a negative pregnancy test (serum or urine) within 7 days prior to treatment.
* (Continuation of # 8) Acceptable contraception includes double-barrier methods (any double combination of: male or female condom with spermicidal gel, diaphragm, sponge, cervical cap, IUD).
* Signed written informed consent document. Written informed consent must be obtained prior to any evaluations being performed solely for the purposes of screening for eligibility for this study.

Exclusion Criteria:

* Prior treatment with any investigational drug within the preceding 2 weeks
* Chronic treatment with systemic steroids or another immunosuppressive agent. Patients can not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Limits for fasting lipids must be: cholesterol </= 300mg/dL and triglyceride </= 2.5 times upper limits of normal (ULN). Patients may be allowed to enroll on the trial after initiation of lipid lowering agents
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases (Brain imaging studies are not required if the patient does not have a history of brain metastases and has no neurological signs or symptoms)
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction </= 6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia; severely impaired lung function (oxygen dependent, Common Terminology Criteria (CTC) Grade 3 or 4 dyspnea); uncontrolled diabetes as defined by fasting serum glucose >1.5 times ULN; any active (acute or chronic) or uncontrolled infection / disorders
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy ; liver disease such as cirrhosis, known chronic active hepatitis or chronic persistent hepatitis; A known history of HIV seropositivity
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 and/or erlotinib (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis (if coumarin is used, weekly monitoring is recommended)
* Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001). Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Acceptable contraception includes double-barrier methods (any double combination of: male or female condom with spermicidal gel, diaphragm, sponge, cervical cap, intrauterine device [IUD]).
* Patients who have received prior treatment with an mTor inhibitor
* Patients with a known hypersensitivity to erlotinib, RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Javle MM, Shroff RT, Xiong H, Varadhachary GA, Fogelman D, Reddy SA, Davis D, Zhang Y, Wolff RA, Abbruzzese JL. Inhibition of the mammalian target of rapamycin (mTOR) in advanced pancreatic cancer: results of two phase II studies. BMC Cancer. 2010 Jul 14;10:368. doi: 10.1186/1471-2407-10-368. PMID 20630061
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2008 through January 20, 2009. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the sixteen registered, one (1) participant was enrolled but did not receive the planned treatment.
Period: Overall Study
Arm/Group | Erlotinib + RAD001
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib + RAD001
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 63 [34 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Surviving at 6 Months
Description: Overall survival (OS) at 6 months in participants receiving a combination of Erlotinib and RAD001 who have received previous treatment for advanced pancreatic cancer. OS at 6 months is number of participants alive at 6 months.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Erlotinib + RAD001
Number analyzed (Participants) | 15
Participants | 15 [34 to 75]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from March 07, 2008 to August 12, 2008 or a total of 6 months.
Arm/Group | Erlotinib + RAD001
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + RAD001 (N=16)
Abdominal Pain (Gastrointestinal disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 7
Alkaline Phosphatase (Metabolism and nutrition disorders) | 5
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Gastrointestinal disorders) | 6
Bilirubin (Metabolism and nutrition disorders) | 1
Cholesterol (serum high) (Metabolism and nutrition disorders) | 1
Confusion (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 3
Dehyration (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 9
Distention/bloating (Gastrointestinal disorders) | 1
Dizziness (General disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Dry eyes (Eye disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Fatigue (General disorders) | 6
Fever without neutropenia (General disorders) | 4
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4
Hypoatremia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Infection with normal neutrophils (Infections and infestations) | 2
Leukocytes (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 5
Mood Alteration (Anxiety) (General disorders) | 2
Mucositis (oral) (Gastrointestinal disorders) | 2
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Pain (back) (Musculoskeletal and connective tissue disorders) | 2
Pain(joint) (Musculoskeletal and connective tissue disorders) | 1
Rash (hand and foot eeaction) (Skin and subcutaneous tissue disorders) | 1
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 2
Rigor/chills (General disorders) | 1
Serum glutamic oxaloacetic transaminase (AST, SGOT) (Metabolism and nutrition disorders) | 2
Serum glutamic pyruvic transaminase (ALT) (Metabolism and nutrition disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 1
Thrombosis (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight Loss (Investigations) | 5
Xerostoma (General disorders) | 1
Yeast infection (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No